CLINICAL TRIAL: NCT07046234
Title: Point of Care Lung Ultrasound Examination in Patients With Shortness of Breath
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Northwestern University (Other); Rush University Medical Center (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SA-000147
Record Dates: First submitted 2025-06-06; First posted 2025-07-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lung Disease; Lung Ultrasound
Keywords: Lung Ultrasound; Artificial Intelligence
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Cohort 1 -Device 1 (Experimental): Cohort 1 will utilize the Vscan Air CL (curvilinear and linear probes) and SL (sector probe) handheld ultrasound to perform an 8-zone lung ultrasound (LUS) exam.
  The Trained HCP will be required to capture at least 2 clips per zone using an ultrasound with Caption AI before moving onto the next zone. The scanner can capture multiple clips per zone, via-auto-capture or Save Best Clip (Study Exam).
  The Expert LUS user will use the same ultrasound system but without Caption Lung AI (Control Exam).
  Interventions: Device: Lung ultrasound
- Cohort 2 -Device 2 (Experimental): Cohort 2 will utilize the Venue GO ultrasound system to perform a 12-zone lung ultrasound (LUS) exam.
  All Qualified users using Caption Lung AI will be required to capture at least 2 clips per zone before moving onto the next zone. The scanner can capture multiple clips per zone, via-auto-capture or Save Best Clip (Study Exam).
  The Qualified user will use the same ultrasound system but without Caption Lung AI (Control Exam).
  Interventions: Device: Lung ultrasound
- Cohort 0 - Vscan (no AI) (Active Comparator): Cohort 0 will utilize the Vscan Air CL (curvilinear and linear probes) and SL (sector probe) handheld ultrasound to perform the following lung ultrasound (LUS) exams.: Each patient will undergo 2 8-zone lung examinations which will be a combination of the enrollment distribution listed below equating to up to 30 subjects with 2 scans per subject (60 scans).
  Interventions: Device: Lung ultrasound

INTERVENTIONS:
Device: Lung ultrasound — Lung ultrasound software.
  Other Names: SaMD

SUMMARY:
This is a prospective, non-randomized clinical validation research study. Subjects will consent and have two ultrasounds as part of the study.

DETAILED DESCRIPTION:
This study is to collect data to validate the performance of Caption Lung AI in enabling trained healthcare professionals to perform LUS to obtain diagnostic-quality Lung Ultrasound Studies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients over the age of 22; AND
* 2. Patients with known lung pathology or patients with no known lung pathology in the hospital or presenting to the hospital or outpatient setting with shortness of breath.

Exclusion Criteria:

* 1. Patients in extremis and/or patients in whom a lung ultrasound would not normally be performed;
* 2. Patients who are unable to consent;
* 3. Patients who are prisoners; AND
* 4. Patients who do not speak English fluently.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: % of patient studies composed of images acquired by the THCPs with sufficient quality to make a clinical assessment | 7 months
  The primary endpoint will be based on the majority assessment of the independent expert readers qualitatively assessment of the LUS exam (study level) as being of diagnostic quality.
Cohort 2: % of patient studies composed of images acquired by the Qualified user to make a clinical assessment | 7 months
  The primary endpoint will be based on the majority assessment of the independent expert readers qualitatively assessment of the LUS exam (study level) as being of diagnostic quality.

SECONDARY OUTCOMES:
Cohort 1: | 7 months
  Sub-group analyses will be performed on the diagnostic image quality performance, with descriptive statistics reported based on age (< 65, ≥ 65), BMI group (< 25, 25 ≤ BMI < 30, ≥ 30), gender (Male / Female), site location, THCP, and zone of the image (1 - 8). The statistical analysis procedure and all applicable performance metrics that were used on the whole sample (i.e., the Primary Outcome Measures) will be repeated for each sub-group level. This will be conducted to ensure that there is no inherent bias where a specific sub-group level has a greater impact on the overall whole-sample performance compared to other levels.
Cohort 2: | 7 months
  Sub-group analyses will be performed on the diagnostic image quality performance, with descriptive statistics reported based on age (< 65, ≥ 65), BMI group (< 25, 25 ≤ BMI < 30, ≥ 30), gender (Male / Female), site location, THCP, and zone of the image (1 -12). The statistical analysis procedure and all applicable performance metrics that were used on the whole sample (i.e., the Primary Outcome Measures) will be repeated for each sub-group level. This will be conducted to ensure that there is no inherent bias where a specific sub-group level has a greater impact on the overall whole-sample performance compared to other levels.
Cohort 1: | 7 months
  Task-based comparison of the study and control exams:
  o Aided non-experts (i.e., THCP) and unaided experts (i.e., Expert LUS user) clips will be reviewed by expert readers for "normal" and "abnormal" ultrasound assessment at the zone level (B-lines, Pleural effusion, Non-aerated Lung / Consolidation, Lung Sliding).
Cohort 2: | 7 months
  Task-based comparison of the study and control exams:
  o Aided user and unaided user (i.e., Qualified user) clips will be reviewed by expert readers for "normal" and "abnormal" ultrasound assessment at the zone level (B-lines, Pleural effusion, Non-aerated Lung / Consolidation, Lung Sliding).
Cohort 1 and 2: | 7 months
  Recording mode (% of clips acquired with auto-capture rate versus save best clip).
Cohort 1: | 7 months
  Acquisition time to complete the LUS exam and for each view (1 - 8).
Cohort 2: | 7 months
  Acquisition time to complete the LUS exam and for each view (1 - 12).
Cohort 1 and 2: | 7 months
  Inter-rater (physician image-interpretation) variability.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Yale University School of Medicine, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Northwestern University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No